CLINICAL TRIAL: NCT06994611
Title: Endoscopic Ultrasound-guided Fine-needle Biopsy With or Without Macroscopic On-site Evaluation for Diagnosis of Solid Pancreatic Lesions: A Prospective Multicenter Randomized Controlled Non-Inferiority Trial
Brief Title: Fine-needle Biopsy Combined With Macroscopic On-site Evaluation for Diagnosis of Solid Pancreatic Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Department of Gastroenterology, Changhai Hospital, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: KTSB20250327028
Record Dates: First submitted 2025-04-28; First posted 2025-05-29 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Diseases
Keywords: EUS-FNB; solid pancreatic lesion; sample processing; 22D Franseen Needle
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MOSE group (Experimental): Patients assigned to this group will receive EUS-FNB as routine. The obtained tissue will be evaluated by Macroscopic On-site Evaluation
  Interventions: Procedure: MOSE application
- Non-mose group (Active Comparator): Patients assigned to this group will receive EUS-FNB as routine. Two needles were punctured and all tissue strips were placed into bottle A formalin.
  Interventions: Procedure: Conventional processing

INTERVENTIONS:
Procedure: MOSE application — The length of the tissue strips was judged using the specimen table and photographed for record. If the MVC of the first needle sample was ≥10mm, the tissue strip was placed into bottle A formalin for fixation. A second needle of tissue strip was pushed directly into the B-bottle formalin. If the first needle sample MVC was < 10mm, the puncture was continued until the total length of sample MVC was ≥10mm, and all samples were placed into bottle A formalin.
  Arms: MOSE group
Procedure: Conventional processing — Two needles were punctured and all tissue strips were placed into bottle A formalin.
  Arms: Non-mose group

SUMMARY:
The goal of this clinical trial is to compare the diagnostic efficacy, core tissue acquisition ability, number of punctures and puncture time of macroscopic on-site evaluation (MOSE) and two punctures alone in Endoscopic ultrasound guided fine-needle biopsy (EUS-FNB) for solid pancreatic lesions. The main questions it aims to answer is: whether the diagnostic accuracy of EUS-FNB performed with two needle passes is not inferior to that of MOSE.

Participants with solid pancreatic lesions who needs histological diagnosis will receive EUS-FNB using 22G Franseen.

In Group 1, the macroscopically visible core (MVC) of the specimen was assessed. If the MVC of the sample obtained from the first needle was ≥10mm, the tissue strip was placed in Bottle A and fixed with formalin. A second needle was then used to obtain another tissue strip, which was directly placed into Bottle B containing formalin. However, if the MVC of the first needle sample was < 10mm, the puncture procedure was continued until the cumulative length of sample's MVC was ≥10mm, and all the sample collected during this process were placed into Bottle A and fixed with formalin. In Group 2, two needles were used to obtain tissue strips, and all the tissue strips were placed into Bottle A formalin.

Researchers will compare the diagnostic efficacy, core tissue acquisition ability, number of punctures and puncture time between the MOSE technique and two-needle puncture method.

ELIGIBILITY:
Inclusion Criteria:

* (Before the trial, subjects must meet all of the requirements listed below in order to be enrolled)

  1. 18-80 years old (inclusive), male and female;
  2. patients with pancreatic solid mass > 1cm detected by CT/MRI/PET-CT or EUS and requiring EUS-FNB diagnosis.
  3. written informed consent was obtained;

Exclusion Criteria:

* (Before the trial, participants could not be enrolled if they met any of the following requirements)

  1. contraindications to endoscopy, such as severe cardiovascular and cerebrovascular diseases;
  2. bleeding coagulation dysfunction (prothrombin international normalized ratio ≥1.5, platelet count ≤ 50 000) or use of antiplatelet drugs;
  3. confirmed pregnancy or possible pregnancy;
  4. pathological diagnosis has been obtained by other methods;
  5. refuse to participate in the study, are participating in another observational clinical trial, or have participated in another clinical trial within 60 days.
  6. other situations where EUS-FNB could not be performed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | 6 months
  Diagnostic accuracy was calculated as the proportion of true positive and true negative in all evaluated cases.

SECONDARY OUTCOMES:
Median puncture number | 2 months
  In the MOSE group, if the MVC of the first needle sample was ≥10mm, an additional needle was inserted. If the MVC of the first stitch is < 10mm, continue to puncture until the total length of the MVC of the sample is ≥10mm. In the non-MOSE group, fixed puncture was performed with 2 needles.
Tissue adequacy | 2 months
  Grade A, existing core tissue (defined as structurally intact tissue with a long axis length of at least 550 μm) that clearly characterizes the lesion and is sufficient for diagnosis; Grade B, the presence of core fragments that do not meet the histological criteria for structural integrity, but can still be diagnosed based on cell morphology; Grade C, no diseased tissue is found and no diagnosis can be made based on the sample.
Puncture time | 2 months
  The puncture time of the MOSE group was defined as the beginning of puncture to the end of the confirmation of sufficient MOSE, and the puncture time of the non-MOSE group was defined as the beginning of puncture to the end of 2 stitches.

OTHER OUTCOMES:
Diagnostic sensitivity | 2 months
  Diagnostic sensitivity was calculated as the proportion of true positives in patient cases.
Diagnostic specificity | 2 months
  Diagnostic specificity was calculated as proportion of true negative in healthy cases.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Shen Li, M.D, Principal Investigator — Department of Gastroenterology, Changhai Hospital, Naval Medical University (Second Military Medical University), shanghai, China
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No